CLINICAL TRIAL: NCT07407621
Title: Effects of Short Isokinetic Eccentric Resistance Training on Neuromuscular Induced Adaptations Among Obese, Untrained Women
Brief Title: Effects of Short Isokinetic Eccentric Resistance Training on Neuromuscular Induced Adaptations
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Nazirah Gulam Mohamed, Mrs, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: USM/JEPeM/PP/24080735
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Physical Inactivity
Keywords: Eccentric; Cardiometabolic; Neuromuscular adaptation
MeSH Terms: conditions — Obesity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECC ISO (Experimental): Eccentric Isokinetic Exercise
  Interventions: Other: ECC ISO
- CON ISO (Active Comparator): Concentric Isokinetic Exercise
  Interventions: Other: CON ISO

INTERVENTIONS:
Other: ECC ISO — Eccentric Isokinetic Exercise
  Arms: ECC ISO
Other: CON ISO — Concentric Isokinetic Exercise
  Arms: CON ISO

SUMMARY:
The study compares the impact of isokinetic resistance training (RT) -induced neuromuscular adaptation following an 8-week short ECC ISO RT and CON ISO RT among obese, untrained women. The main question it aims to answer is:

1. Does exercise-induced neuromuscular adaptation following progressive short ECC ISO RT, more effectively than CON ISO RT, among obese, untrained women?

Researchers will compare drug ECCISO RT to a CONISO RT to see if ECCISO RT is more effective in inducing neuro-muscular adaptations in obese, untrained women.

Participants will:

1. Train on isokinetic ECC or CON for 8 weeks
2. Visit the clinic twice for baseline and post tests

DETAILED DESCRIPTION:
1.1 Introduction

Exercise-induced neuromuscular and functional changes are mode-specific. Exercise-induced muscular adaptations may be influenced by mechanical tension, subcellular damage, and metabolic stress. Eccentric (ECC) contraction happens when the external force exerted on the muscle exceeds the momentary force generated by the muscle. As a result, the muscle's strength is sufficient to overcome the load or resistance that causes the muscle to lengthen. Compared with concentric (CON) or isometric (ISO) contractions, ECC training elicits greater mechanical strain and microlesions in the muscles, which may lead to more pronounced muscular adaptations. ECC exercise is traditionally performed against a constant external load or at a constant velocity (isokinetic). Depending on the type of training, this produces varying mechanical demands, resulting in distinct neuromuscular and muscle-tendon adaptation mechanisms. In contrast to ISO or CON muscular contractions, the central nervous system employs a distinct neural strategy to govern skeletal muscle contraction. Different activation levels among synergistic muscles during ECC contractions compared with CON contractions, and the preferential recruitment of rapid-twitch motor units, are two examples of how this is demonstrated.

1.2 Problem statement & study rationale

Emerging data suggest that adiposity is associated with muscular weakness and reduced muscle quality. Regular resistance training (RT) has been shown to enhance a muscle's maximal regenerative capacity. It is believed that neural mechanisms primarily contribute to the initial (<2-4 weeks) gains in muscle force production during resistance training, followed by adaptations in muscle morphology (>5-8 weeks). However, this evidence is based on combining both ECC and CON contraction exercises. Studies have shown that ECC contraction elicits greater neuromuscular adaptation than CON contraction. Therefore, ECC RT is a promising approach for individuals with muscular weakness, such as the obese. Hence, it is postulated that short progressive eccentric isokinetic resistance training (ECCISO RT) will increase neuromuscular adaptations in obese untrained women compared to concentric isokinetic resistance training (CONISO RT)

2.0 Literature Review

2.1 Introduction

The higher prevalence of musculoskeletal pain, mechanical loading, poor muscle fitness, and other musculoskeletal problems is linked to obesity. The flexors and extensors of the lower limbs are responsible for balance, mobility, and the ability to perform daily tasks. The strength and endurance of skeletal muscles are altered by excess fat mass (FM). The amount of muscle in the mid-thigh is roughly 2.5 times that of fat mass; however, obese people have more intra- and intermuscular fat, fat between muscle cells, which has a detrimental effect on force production and functional independence. The force-producing ability of a skeletal muscle can be used to evaluate the muscle's functional capacity. The ability to apply force, one's absolute strength, is necessary to carry out daily tasks. Obese people have been shown to have higher absolute maximum voluntary contraction (MVC) torques than normal-weight people. Nevertheless, they also have lower muscle strength relative to body weight and fat-free mass (FFM).

2.2 The impact of obesity on skeletal muscle composition and strength

Although total muscle mass is higher in overweight and obese individuals, the relative muscle strength of overweight and obese people is significantly lower than that of healthy people, which can lead to a decrease in physical function. Obesity can increase the absolute force and power of the weight-bearing muscles in the lower extremities due to increased demand (Marte Johannson, 2021). However, when force production and power output are normalized to total body mass, a decline is observed with higher BMI, resulting in reduced muscle quality and fatigue resistance. Moreover, the negative impact of adipose tissue-dependent metabolic adaptations, such as oxidative stress, inflammation, and insulin resistance, harms muscle mass metabolism.

The proportion of muscle fibres differs in obese individuals. A positive association exists between body fatness and the type II muscle fibre ratio, with higher type IIX fibre content reported in overweight individuals. Type II muscle fibres often have lesser numbers of mitochondria, myoglobin, and capillaries than slow-twitch fibres, making them more susceptible to tiredness. Type IIX (also known as Type IIB) fibres generate the maximum force; however, they are highly inefficient due to their high myosin ATPase activity, low oxidative capacity, and dependency on anaerobic metabolism. Type IIA fibres, commonly called intermediate muscle fibres, combine type I and IIX fibres with equivalent tension. These fibres, which can use both aerobic and anaerobic energy sources, have greater oxidative capacity and fatigue more slowly than type IIX fibres. An increased proportion of type II muscle is associated with increased (a) insulin resistance, (b) risk of hyperinsulinemia, (c) decreased fatigue resistance/exercise tolerance, (d) endurance, and (e) mobility.

Both human and animal studies have found that Type II (particularly IIx) muscle fibres are more susceptible to injury following ECC activity -increased type IIx fibres and sedentarism are associated with greater muscle damage among overweight individuals with ECC training. A single bout of high-force ECC exercise increases muscle fibre Satellite cells (SCs) content and activation status in Type II. SCs are essential in skeletal muscle tissue growth, repair, and regeneration. Hence, ECC training is a promising exercise technique for individuals with physical function limitations, including overweight and obese individuals.

2.3 Effects of eccentric resistance training on neuromuscular adaptation

Compared with traditional (CON) exercise, ECC exercise training significantly increases muscular strength. Muscle strength gains in ECC training are likely attributable to a combination of neurological, morphological, and anatomical factors. Studies have shown that ECC contraction elicits greater neuromuscular adaptation than CON contraction. Although a recent meta-analysis found no statistically significant differences in strength gains between ECC and CON training, ECC exercise training also showed a trend toward greater improvements in CON strength than CON exercise. This demonstrates the mode-specificity of the neuromuscular and functional adaptations caused by ECC exercise. ECC training has increased surface electromyographic (EMG) activity during contractions but not during CON contractions. However, conflicting outcomes have been reported. The electrical stimulation of muscle is thought to be represented by the maximal EMG (i.e., peak root mean square [RMS] values and integrated voltage from the EMG [iEMG]) after training (Douglas et al., 2017). This is influenced by the quantity and size (i.e., type I vs type II fibres) of recruited motor units, motor unit discharge rate, and motor unit synchrony.

Several studies have found that ECC RT improves muscle power, as measured primarily by lower-body jump variants. Healthy, trained men (N=24) were randomly assigned to groups: ECC RT (n=12) and CON RT (n=12). The quadriceps' maximal voluntary isometric contraction (MVCISO), vertical jumping, and multichannel surface EMG signals were measured pre- and post-RT. Raw EMG signals were used to calculate muscle fibre conduction velocity (MFCV) and root mean square (RMS). Following ECC RT, there was a statistically significant increase in vertical jumping and MVCISO percentages compared to CON RT. Similarly, ECC RT increased EMG MFCV and RMS more than concentric exercise.

Twenty healthy male subjects underwent 12 weeks of ECCISO RT on an isokinetic dynamometer, and neuromuscular evaluations of the knee extensors were performed every 4 weeks. The ECCISO RT comprised 3 sets of 10 repetitions during weeks 1-4, 4 sets in weeks 5-8, and 5 sets in weeks 9-12. A 1-minute rest period was respected between sets. Significant improvements were observed in muscular strength [PTECC (29 %), PTISO (24 %) & PTCON (15 %)], electromyographic activity [ΣEMGECC (33 %), EMGISO (29 %)] and muscle mass [Knee extensor muscle thickness (ΣMT 10 %) and anatomical rectus femoris anatomical cross-sectional area (ACSA rf 19 %)] post-training. ECC and ISO activation increased at 4 and 8 training weeks, respectively, whereas CON activation did not change. These findings imply that the proportional increase in neuronal activation and muscle mass accounts for ECC and ISO strength gains through 8 training weeks, whereas other processes appear to be involved in the increments in the final 4 training weeks. Meanwhile, the relative increase in PTCON was negligible and unrelated to neural adaptation following ECCISO RT.

Synergistic muscles exhibit distinct morphological and neurophysiological adaptations in response to ECCISO RT. Healthy males (N=20) were assessed for neural and muscular adaptation in vastus medialis (VM) and vastus lateralis (VL) following progressive ECCISO RT for 12 weeks. Morphological and neural adaptations were evaluated using ultrasound measurements of VL and VM muscle thickness at rest and electromyographic measurements during MVCISO. Post-training, the thickness of both muscles increased significantly (VL: 6.9%; VM: 15.8%). However, there were significant increases in muscle activity in VM (47.8%; p =.003) but not in VL (19.8%).

2.4 Conclusion

The early adverse effects of eccentric exercise include subcellular muscle injury, discomfort, decreased fibre excitability, and initial muscular weakening. An effective stimulus for eliciting physiological and neuronal training responses is stretch and overload, as in eccentric contractions. Enhancement in muscle function results from adaptations induced by eccentric exercise, including muscle growth, increased cortical activity, and modifications in motor unit behaviour.

ELIGIBILITY:
INCLUSION CRITERIA:

* Eumenorrheic women (reporting menstrual cycle between 21-35 days)
* Age 25-45 y/o
* BMI > 23.0 kg/m2
* Body fat percentage > 30%
* No lower limb orthopaedic injuries
* Have not participated in any structured/ unstructured weight loss intervention in the past 12 months
* Sedentary lifestyle (regular exercise <1 hour per week)
* Stable body weight (loss or gain of no greater than 2 kg)
* Stable medication use for six months before enrolment

EXCLUSION CRITERIA:

* smokers
* taking supplements or medication known to affect REE (such as oral contraceptives)
* severe medical conditions affecting their physical or mental health
* individuals with an implanted medical device
* suffer from alcohol or drug abuse
* trying to conceive/ pregnant, or breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximal voluntary strength | 8 weeks
  Changes in maximal voluntary strength
Neural activation assessment | 8 weeks
  Changes in neural activation during strength
Fasting plasma glucose | 8 weeks
  Changes in fasting plasma glucose
Functional physical fitness (6-minute walking test) | 8 weeks
  Changes in distance during 6-minute walking test
Indirect calorimetry | 8 weeks
  Changes in basal metobolic rate/ fat oxidation rate/ charbohydrate oxidation rate
HDL cholesterol | 8-weeks
  Changes in HDL cholesterol
LDL cholesterol | 8-weeks
  Changes in LDL cholesterol
Total cholesterol | 8-weeks
  Changes in total cholesterol
Trigliceride | 8-weeks
  Changes in triglyceride

SECONDARY OUTCOMES:
Percentage of Body Fat | 8 weeks
  Changes in the percentage segmental of body fat
Lean muscle mass | 8 weeks
  Percentage of changes in segmental ean muscle mass

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Munir Che Muhamed, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Department of Community Health, Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peñailillo, L., Diaz-Reiher, M., Gurovich, A. and Flores-Opazo, M., 2022. A Short-Term Eccentric HIIT Induced Greater Reduction in Cardio-Metabolic Risk Markers in Comparison With Concentric HIIT in Sedentary Overweight Men. Research Quarterly for Exercise and Sport [online]. Available from: https://www.tandfonline.com/action/journalInformation?journalCode=urqe20.
- [Background] Paschalis, V., Nikolaidis, M. G., Theodorou, A. A., Panayiotou, G., Fatouros, I. G., Koutedakis, Y. and Jamurtas, A. Z., 2011. A Weekly Bout of Eccentric Exercise Is Sufficient to Induce Health-Promoting Effects. Medicine & Science in Sports Exercise [online], 43 (1), 64-73. Available from: http://www.acsm-msse.org [Accessed 19 Apr 2022].
- [Background] Julian, V., Thivel, D., Miguet, M., Pereira, B., Costes, F., Coudeyre, E., Duclos, M. and Richard, R., 2019. Eccentric cycling is more efficient in reducing fat mass than concentric cycling in adolescents with obesity. Scandinavian Journal of Medicine & Science in Sports [online], 29 (1), 4-15. Available from: https://onlinelibrary.wiley.com/doi/full/10.1111/sms.13301 [Accessed 19 Apr 2022].
- [Background] Pereira, B., Perrault, H., Duclos, M. and Richard, R., 2018. Eccentric Training Improves Body Composition by Inducing Mechanical and Metabolic Adaptations: A Promising Approach for Overweight and Obese Individuals. Frontiers in Physiology | www.frontiersin.org [online], 1, 1013. Available from: www.frontiersin.org.
- [Background] Jeon, S., Ye, X., Miller, W. M. and Song, J. S., 2022. Effect of repeated eccentric exercise on muscle damage markers and motor unit control strategies in arm and hand muscle. Sports Medicine and Health Science, 4 (1), 44-53.
- [Background] Coratella, G., Bollinger, L., Yan, X., Su, H., Liu, X., Gao, Y., Lu, J., Ma, Q., Shi, Y., Liu, J. and Xin, S., 2022. Effects of Different Resistance Exercise Forms on Body Composition and Muscle Strength in Overweight and/or Obese Individuals: A Systematic Review and Meta-Analysis. Frontiers in Physiology | www.frontiersin.org [online], 12, 791999. Available from: www.frontiersin.org.
- [Background] Chen, T. C., Hsieh, C.-C., Tseng, K.-W., Ho, C.-C. and Nosaka, K., 2017. Effects of Descending Stair Walking on Health and Fitness of Elderly Obese Women. Medicine and science in sports and exercise, 49 (8), 1614-1622.